CLINICAL TRIAL: NCT06390280
Title: The Role of High Intraoperative Fraction of Inspired Oxygen in Preventing Postoperative Nausea and Vomiting in Laparoscopic Cholecystectomy
Brief Title: The Role of High Intraoperative Fraction of Inspired Oxygen in Preventing Postoperative Nausea and Vomiting
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Zeynep sym, Principal Investigator, Ankara City Hospital Bilkent
Other Study IDs: E2-22-2167
Record Dates: First submitted 2023-11-14; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Nausea and Vomiting; Laparoscopic Cholecystectomy
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- grup I: Intraoperative Fraction of Inspired Oxygen %30 applied
  Interventions: Procedure: intraoperative Fraction of Inspired Oxygen
- grup II: Intraoperative Fraction of Inspired Oxygen %80 applied
  Interventions: Procedure: intraoperative Fraction of Inspired Oxygen

INTERVENTIONS:
Procedure: intraoperative Fraction of Inspired Oxygen — Group I intraoperative Fraction of Inspired Oxygen 30%, Group II intraoperative Fraction of Inspired Oxygen 80% applied group.

SUMMARY:
Postoperative nausea and vomiting is one of the most common complications after laparoscopic surgeries.

The investigators aimed to evaluate the effects of intraoperative high fraction of inspired oxygen in preventing postoperative nausea and vomiting according to Apfel score in laparoscopic cholecystectomy patients.

DETAILED DESCRIPTION:
All participants will be monitored with electrocardiogram, pulse oximeter , non-invasive blood pressure. The fasting period of the patients was 8 hours. The participants were randomly divided into two groups by the auxiliary health personnel using the closed envelope draw method. After the participants were taken to the operating room, their files were checked, consent for the study was obtained, and the Apfel score was noted. Participants were started on intravenous crystalloid fluid infusion at 8ml/kg/hour. After induction of general anesthesia with 0.03mg/kg midazolam, 2-2.5 mg/kg propofol, 1 µg/kg remifentanil, 0.6 mg/kg rocuronium, the participants were intubated and connected to the anesthesia machine, with sevoflurane and maintenance administered at minimum alveolar concentration 1.3. was achieved with remifentanil infusion. After the participants were connected to the anesthesia device, the tidal volume was adjusted to 7 ml/kg, respiratory rate 12-14/min, positive end-expiratory pressure 5 cmH2O, flow 2 liter/min, Fraction of inspired oxygen 30% in Group I and 80% in Group 2. Gastric fluid and air were aspirated from the participants using an orogastric tube. The participants' vitals were monitored intraoperatively at 5-minute intervals and recorded every 15 minutes. Intra-abdominal pressure was kept between 10-12 mmHg. Approximately 15 minutes before the end of the surgical procedure, remifentanil infusion was stopped, and 1 g paracetamol and 50 mg dexketoprofen i.v. were administered as postoperative analgesics was given. No narcotic analgesics were given. At the end of the operation, exsufflation was performed before the trocars were removed and the intra-abdominal pressure was allowed to return to normal. The surgical team was given bupivacaine to administer 15 mg per trocar site. While the last few skin stitches were being placed, sevoflurane was discontinued in all participants and they were switched to 100% oxygen. Muscle relaxant antagonism was achieved with sugammadex (2 mg/kg) in both groups. The patients were extubated and monitored for 1 hour postoperatively in the recovery unit. All patients were given 2 liter/min O2 in the recovery unit. In case of nausea and vomiting, the Nausea Vomiting Score is noted and 4 mg of ondansetron i.v. is given to patients with moderate to severe nausea and vomiting. Participants requiring additional analgesics were given 100 mg tramadol. Postoperative 24-hour nausea and vomiting was monitored in the patient's hospitalization ward. The participants with nausea and vomiting during the 24-hour follow-up were learned from the follow-up doctor and noted on the follow-up forms. During the ward follow-up, patients with nausea were given 4mg of ondansetron.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective laparoscopy cholecystectomy surgery
* Patients younger than 60 years old
* Both genders
* American Society of Anesthesiologists (ASA) I-II risk group

Exclusion Criteria:

* pregnancy, patients who do not want to participate in the study, surgery time > 2 hours

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A total of 98 patients, under the age of 60, in the ASA I-II risk group, who underwent laparoscopic cholecystectomy surgery were included.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2022-07-10 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting | at the postoperative 15.minutes
  the investigators aimed to compare postoperative nause and vomiting
Postoperative nausea and vomiting 24.hours | at the postoperative 24.hours
  the investigators aimed to compare postoperative nause and vomiting

SECONDARY OUTCOMES:
Postoperative antiemetic 15. minutes | at the postoperative 15.minutes
  the investigators aimed to compare postoperative making antiemetic medication
Postoperative antiemetic 24.hours | at the postoperative 24.hours
  the investigators aimed to compare postoperative making antiemetic medication

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Bilkent, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided